CLINICAL TRIAL: NCT02453438
Title: Mood Patient Powered Research Network (MoodNetwork)
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Andrew A. Nierenberg, MD, Director, Bipolar Clinic and Research Program, Massachusetts General Hospital
Other Study IDs: 2014P001346
Record Dates: First submitted 2015-05-05; First posted 2015-05-25 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Mood Disorders; Bipolar Disorder; Major Depressive Disorder; Depression
MeSH Terms: conditions — Mood Disorders; Bipolar Disorder; Depressive Disorder, Major; Depression | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Patient Reported Outcomes — Patient reported outcomes will be collected using a variety of questionnaires that assess mood symptoms.

SUMMARY:
The MoodNetwork, a patient-powered research network (PPRN), is one of 18 PPRNs participating in Patient-Centered Outcomes Research Institute's (PCORI) PCORnet network. Its objective is to improve the nation's capacity to conduct comparative effectiveness research that reflects questions of greatest importance to patients and other stakeholders. A robust data infrastructure will be built that, in phase one, allows participants to contribute data, including those from participant questionnaires, visualize their own health information in intuitive and helpful ways, and share their aggregated de-identified health information within and outside of the Network.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Valid email address
* Self-identify as having a mood disorder

Exclusion Criteria:

* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: English speaking individuals over 18 years of age who self-identify as having a mood disorder.
Sampling Method: Non-Probability Sample
Enrollment: 5716 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Patient Reported Outcomes Working Group Items Questionnaire | average of 3 years
Composite International Diagnostic Interview Mania Questionnaire | average of 3 years
Mini International Neuropsychiatric Interview Depression | average of 3 years
Quick Inventory of Depressive Symptoms Self Report | average of 3 years
Altman Self Rated Mania Scale | average of 3 years
WHO-five well-being index (WHO-5) | average of 3 years
Depression and Bipolar Support Alliance Wellness Tracker Questionnaire | average of 3 years
Experience of Care and Health Outcomes Questionnaire | average of 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrew A Nierenberg, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Bipolar Clinic and Research Program, Boston, Massachusetts, United States